CLINICAL TRIAL: NCT02544074
Title: Validity of the Electronic Self-Administered Gerocognitive Examination (eSAGE)
Acronym: eSAGE
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Brain Test, Inc. (Industry)
Responsible Party: Principal Investigator, Douglas Scharre, Professor, Ohio State University
Other Study IDs: 2014H0039
Record Dates: First submitted 2015-03-18; First posted 2015-09-09 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Mild Cognitive Impairment; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (31):
- eSAGE score of 10: Participants who score a 10 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 11: Participants who score an 11 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 12: Participants who score a 12 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 13: Participants who score a 13 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 14: Participants who score a 14 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 15: Participants who score a 15 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 16: Participants who score a 16 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 17: Participants who score a 17 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 18: Participants who score a 18 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 19: Participants who score a 19 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 20: Participants who score a 20 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 21: Participants who score a 21 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 22: Participants who score a 22 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 9: Participants who score a 9 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 8: Participants who score an 8 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 6: Participants who score a 6 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 7: Participants who score a 7 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 5: Participants who score a 5 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 4: Participants who score a 4 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 3: Participants who score a 3 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- eSAGE score of 2: Participants who score a 2 on the eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: neuropsychological testing
- Smartphone eSAGE score of 13: Participants who score a 13 on the smartphone eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: eSAGE testing
- Smartphone eSAGE score of 14: Participants who score a 14 on the smartphone eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: eSAGE testing
- Smartphone eSAGE score of 15: Participants who score a 15 on the smartphone eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: eSAGE testing
- Smartphone eSAGE score of 16: Participants who score a 16 on the smartphone eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: eSAGE testing
- Smartphone eSAGE score of 17: Participants who score a 17 on the smartphone eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: eSAGE testing
- Smartphone eSAGE score of 18: Participants who score a 18 on the smartphone eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: eSAGE testing
- Smartphone eSAGE score of 19: Participants who score a 19 on the smartphone eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: eSAGE testing
- Smartphone eSAGE score of 20: Participants who score a 20 on the smartphone eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: eSAGE testing
- Smartphone eSAGE score of 21: Participants who score a 21 on the smartphone eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: eSAGE testing
- Smartphone eSAGE score of 22: Participants who score a 22 on the smartphone eSAGE. Interventions include neuropsychological testing.
  Interventions: Behavioral: eSAGE testing

INTERVENTIONS:
Behavioral: neuropsychological testing — standard neuropsychological testing including brief standardized assessments
  Groups: eSAGE score of 10; eSAGE score of 11; eSAGE score of 12; eSAGE score of 13; eSAGE score of 14; eSAGE score of 15; eSAGE score of 16; eSAGE score of 17; eSAGE score of 18; eSAGE score of 19; eSAGE score of 2; eSAGE score of 20; eSAGE score of 21; eSAGE score of 22; eSAGE score of 3; eSAGE score of 4; eSAGE score of 5; eSAGE score of 6; eSAGE score of 7; eSAGE score of 8; eSAGE score of 9
Behavioral: eSAGE testing — Neuropsychological testing including the eSAGE tablet and eSAGE smartphone
  Groups: Smartphone eSAGE score of 13; Smartphone eSAGE score of 14; Smartphone eSAGE score of 15; Smartphone eSAGE score of 16; Smartphone eSAGE score of 17; Smartphone eSAGE score of 18; Smartphone eSAGE score of 19; Smartphone eSAGE score of 20; Smartphone eSAGE score of 21; Smartphone eSAGE score of 22

SUMMARY:
The Self-Administered Gerocognitive Examination (SAGE) is a valid and reliable cognitive assessment tool used to identify both Mild Cognitive Impairment (MCI) and early dementia. SAGE's self-administered feature, pen and paper format, and four equivalent interchangeable forms allows it to be given in almost any setting, does not require any staff time to administer and makes it practical to rapidly screen large numbers of individuals in the community or in their home.This trial is being conducted to study the validity of SAGE in a digital format (eSAGE) for cognitive screening.

The investigators will analyze the data to learn the correlations between eSAGE and gold standard neuropsychological testing designed to differentiate normal cognition from MCI and early dementia. The investigators will also find out whether the paper (SAGE) and electronic (eSAGE) versions of SAGE could be used interchangeably or not.

Addendum:

The eSAGE was previously validated in an earlier stage of this trial. It was initially designed for tablet use and the exact same test has recently been formatted for smartphone use.

This addendum is being conducted to study the validity of the smartphone eSAGE compared to the tablet eSAGE for cognitive screening.

DETAILED DESCRIPTION:
Participants will be recruited based on their eSAGE scores and evaluated with neuropsychological testing and medical history to determine their status as normal, mild cognitive impairment, or dementia.

The investigators will analyze the data to learn the correlations between eSAGE and gold standard neuropsychological testing designed to differentiate normal cognition from MCI and early dementia. The investigators will also find out whether the paper (SAGE) and electronic (eSAGE) versions of SAGE could be used interchangeably or not.

Addendum:

Subjects will be scheduled for a one time visit where they will be administered both the tablet eSAGE and the smartphone eSAGE. eSAGE tablet scores will be compared to eSAGE smartphone scores to determine if the two formats are equivalent to each other.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 49 years old of either gender
* Vision and hearing sufficient for compliance with tests

Exclusion Criteria:

* Diagnosis by a physician of moderate or severe dementia
* Intellectual disability

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from a wide variety of community events including senior centers, health fairs, educational talks to lay public, independent and assisted living facilities, and free memory screens as well as from ambulatory Geriatric or Memory Disorders Clinics. The SAGE cognitive screening tool will be given to all subjects willing to take the test.Participants who complete the SAGE test and meet inclusion and exclusion criteria will be divided into groups based on their initial SAGE scores. Each group will be composed of subjects with the same score. Individuals will be randomly selected from each group and asked to further participate in a one-time clinical evaluation.
  Addendum:
  Subjects will be recruited from community events and our clinic and research center.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Scharre, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Scharre DW, Chang SI, Nagaraja HN, Vrettos NE, Bornstein RA. Digitally translated Self-Administered Gerocognitive Examination (eSAGE): relationship with its validated paper version, neuropsychological evaluations, and clinical assessments. Alzheimers Res Ther. 2017 Jun 27;9(1):44. doi: 10.1186/s13195-017-0269-3. PMID 28655351

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The eSAGE test is scored from 0-22 with 22 indicating a perfect score.
Period: Overall Study
Arm/Group | eSAGE Score of 2 | eSAGE Score of 3 | eSAGE Score of 4 | eSAGE Score of 5 | eSAGE Score of 6 | eSAGE Score of 7 | eSAGE Score of 8 | eSAGE Score of 9 | eSAGE Score of 10 | eSAGE Score of 11 | eSAGE Score of 12 | eSAGE Score of 13 | eSAGE Score of 14 | eSAGE Score of 15 | eSAGE Score of 16 | eSAGE Score of 17 | eSAGE Score of 18 | eSAGE Score of 19 | eSAGE Score of 20 | eSAGE Score of 21 | eSAGE Score of 22
Started | 1 | 1 | 1 | 1 | 4 | 1 | 2 | 4 | 6 | 2 | 2 | 3 | 4 | 5 | 5 | 8 | 6 | 3 | 4 | 3 | 3
Completed | 1 | 0 | 1 | 1 | 4 | 0 | 2 | 4 | 6 | 1 | 2 | 3 | 4 | 5 | 5 | 8 | 6 | 3 | 4 | 3 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Tablet error | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | eSAGE Score of 2 | eSAGE Score of 3 | eSAGE Score of 4 | eSAGE Score of 5 | eSAGE Score of 6 | eSAGE Score of 7 | eSAGE Score of 8 | eSAGE Score of 9 | eSAGE Score of 10 | eSAGE Score of 11 | eSAGE Score of 12 | eSAGE Score of 13 | eSAGE Score of 14 | eSAGE Score of 15 | eSAGE Score of 16 | eSAGE Score of 17 | eSAGE Score of 18 | eSAGE Score of 19 | eSAGE Score of 20 | eSAGE Score of 21 | eSAGE Score of 22 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 1 | 2 | 4 | 6 | 2 | 2 | 3 | 4 | 5 | 5 | 8 | 6 | 3 | 4 | 3 | 3 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 6
  >=65 years | 1 | 1 | 1 | 1 | 4 | 1 | 2 | 4 | 6 | 2 | 2 | 3 | 4 | 4 | 4 | 5 | 6 | 3 | 4 | 3 | 2 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 3 | 4 | 1 | 2 | 2 | 2 | 4 | 2 | 7 | 3 | 2 | 3 | 2 | 3 | 44
  Male | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 3 | 1 | 3 | 1 | 1 | 1 | 0 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 5
  White | 1 | 1 | 1 | 1 | 3 | 1 | 2 | 3 | 6 | 2 | 2 | 3 | 4 | 2 | 4 | 7 | 6 | 2 | 3 | 3 | 3 | 60
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: eSAGE Score Compared to the Sum of the Neuropsychological Measures.
Description: Analysis will consist of comparing the subject's scores on the SAGE in digital format to their neuropsychological test scores. This will be a composite score of the neuropsychological testing scores. The neuropsychological measures include:
  * Boston Naming Test
  * Wisconsin Card Sort Task (WCST)
  * Hopkins Verbal Learning Test (HVLT)
  * FAS verbal fluency task
  * Wechsler Adult Intelligence Scale III (WAIS III) Letter-number and block design subtests
  Associations will be investigated using Spearman correlations.
Time Frame: 3 Hours
Measure: Number; unit: spearman rank correlation
Groups:
- eSAGE Score Compared to the Sum of Neuropsychological Measures: Analysis will consist of comparing the subject's scores on the SAGE in digital format to their neuropsychological test scores. This will be a composite score of the neuropsychological testing scores. The neuropsychological measures include:
  * Boston Naming Test
  * Wisconsin Card Sort Task (WCST)
  * Hopkins Verbal Learning Test (HVLT)
  * FAS verbal fluency task
  * Wechsler Adult Intelligence Scale III (WAIS III) Letter-number and block design subtests
  Associations will be investigated using Spearman correlations.
Arm/Group | eSAGE Score Compared to the Sum of Neuropsychological Measures
Number analyzed (Participants) | 66
spearman rank correlation | 0.7292

2. Secondary Outcome: eSAGE Score Compared to the Paper SAGE Score
Description: The investigators will compare the subject's scores on the SAGE in digital format to their paper SAGE scores to determine if these two formats are equivalent to each other. Associations will be investigated using Spearman correlations.
Time Frame: 3 hours
Measure: Number; unit: spearman rank correlation
Groups:
- eSAGE Score Compared to the Paper SAGE Score: The investigators will compare the subject's scores on the SAGE in digital format to their paper SAGE scores to determine if these two formats are equivalent to each other. Associations will be investigated using Spearman correlations.
Arm/Group | eSAGE Score Compared to the Paper SAGE Score
Number analyzed (Participants) | 66
spearman rank correlation | 0.8824

3. Secondary Outcome: eSAGE Score Compared to the Mini-Mental State Examination (MMSE) Score
Description: The investigators will compare the eSAGE scores with the Mini-Mental State Examination (MMSE) scores. Associations will be investigated using Spearman correlations.
Time Frame: 3 hours
Measure: Number; unit: spearman rank correlation
Groups:
- eSAGE Score Compared to the Mini-Mental State Exam Score: The investigators will compare the eSAGE scores with the Mini-Mental State Examination (MMSE) scores. Associations will be investigated using Spearman correlations.
Arm/Group | eSAGE Score Compared to the Mini-Mental State Exam Score
Number analyzed (Participants) | 66
spearman rank correlation | 0.6711

4. Secondary Outcome: eSAGE Score Compared to the Montreal Cognitive Assessment (MoCA) Score
Description: The investigators will compare the eSAGE scores with the Montreal Cognitive Assessment (MoCA) scores. Associations will be investigated using Spearman correlations.
Time Frame: 3 hours
Measure: Number; unit: spearman rank correlation
Groups:
- eSAGE Score Compared to the MoCA Score: The investigators will compare the eSAGE scores with the Montreal Cognitive Assessment (MoCA) scores. Associations will be investigated using Spearman correlations.
Arm/Group | eSAGE Score Compared to the MoCA Score
Number analyzed (Participants) | 66
spearman rank correlation | 0.7577

5. Secondary Outcome: eSAGE Score Compared to the Boston Naming Test Score
Description: The investigators will compare the eSAGE scores to the Boston Naming Test score. The Boston Naming Test consists of 60 pictures of nouns that subjects must try to name. Associations will be investigated using Spearman correlations.
Time Frame: 3 hours
Measure: Number; unit: spearman rank correlation
Groups:
- eSAGE Score Compared to the Boston Naming Test Score: The investigators will compare the eSAGE scores to the Boston Naming Test scores. Associations will be investigated using Spearman correlations.
Arm/Group | eSAGE Score Compared to the Boston Naming Test Score
Number analyzed (Participants) | 66
spearman rank correlation | 0.3487

6. Secondary Outcome: eSAGE Score Compared to the Wisconsin Card Sort Task (WCST) Score
Description: The investigators will compare the eSAGE scores to the Wisconsin Card Sort Task (WCST) perseverative errors scores. Associations will be investigated using Spearman correlations.
Time Frame: 3 hours
Measure: Number; unit: spearman rank correlation
Groups:
- eSAGE Score Compared to the WCST Score: The investigators will compare the eSAGE scores to the Wisconsin Card Sort Task (WCST) perseverative errors scores. Associations will be investigated using Spearman correlations.
Arm/Group | eSAGE Score Compared to the WCST Score
Number analyzed (Participants) | 66
spearman rank correlation | 0.4596

7. Secondary Outcome: eSAGE Score Compared to the Hopkins Verbal Learning Test (HVLT) Score
Description: The investigators will compare the eSAGE scores to the Hopkins Verbal Learning Test (HVLT) total learning scores. Associations will be investigated using Spearman correlations. The investigators will also compare the eSAGE scores to the Hopkins Verbal Learning Test (HVLT) delayed recall scores. Associations will be investigated using Spearman correlations.
Time Frame: 3 hours
Measure: Number; unit: spearman rank correlation
Groups:
- eSAGE Score Compared to the HVLT Total Learning Score: The investigators will compare the eSAGE scores to the Hopkins Verbal Learning Test (HVLT) total learning scores. Associations will be investigated using Spearman correlations.
- eSAGE Score Compared to the HVLT Delayed Recall Score: The investigators will compare the eSAGE scores to the Hopkins Verbal Learning Test (HVLT) delayed recall scores. Associations will be investigated using Spearman correlations.
Arm/Group | eSAGE Score Compared to the HVLT Total Learning Score | eSAGE Score Compared to the HVLT Delayed Recall Score
Number analyzed (Participants) | 66 | 66
spearman rank correlation | 0.6045 | 0.4866

8. Secondary Outcome: eSAGE Score Compare to the FAS Verbal Fluency Task Score
Description: The investigators will compare the eSAGE scores to the FAS Verbal Fluency Task scores. Associations will be investigated using Spearman correlations.
Time Frame: 3 hours
Measure: Number; unit: spearman rank correlation
Groups:
- eSAGE Score Compared to the FAS Verbal Fluency Task Score: The investigators will compare the eSAGE scores to the FAS Verbal Fluency Task scores. Associations will be investigated using Spearman correlations.
Arm/Group | eSAGE Score Compared to the FAS Verbal Fluency Task Score
Number analyzed (Participants) | 66
spearman rank correlation | 0.3210

9. Secondary Outcome: eSAGE Score Compared to the Wechsler Adult Intelligence Scale III (WAIS III) Letter-number Score
Description: The investigators will compare the eSAGE scores to the WAIS III Letter-number scores. The WAIS III Letter-number test asks subjects to recall a series of numbers in increasing order and letters in alphabetical order. Associations will be investigated using Spearman correlations.
Time Frame: 3 hours
Measure: Number; unit: spearman rank correlation
Groups:
- eSAGE Score Compared to the WAIS III Letter-number Score: The investigators will compare the eSAGE scores to the WAIS III Letter-number scores. Associations will be investigated using Spearman correlations.
Arm/Group | eSAGE Score Compared to the WAIS III Letter-number Score
Number analyzed (Participants) | 66
spearman rank correlation | 0.5349

10. Secondary Outcome: eSAGE Score Compared to the Wechsler Adult Intelligence Scale III (WAIS III) Block Design Score
Description: The investigators will compare the eSAGE scores to the WAIS III Block Design scores. The WAIS III Block Design requires the replication of red and white designs using three-dimensional colored blocks. Associations will be investigated using Spearman correlations.
Time Frame: 3 hours
Measure: Number; unit: spearman rank correlation
Groups:
- eSAGE Score Compared to the WAIS III Block Design Score: The investigators will compare the eSAGE scores to the WAIS III Block Design scores. Associations will be investigated using Spearman correlations.
Arm/Group | eSAGE Score Compared to the WAIS III Block Design Score
Number analyzed (Participants) | 66
spearman rank correlation | 0.5774

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 1 day, the day of the study visit.
Arm/Group | eSAGE Score of 2 | eSAGE Score of 3 | eSAGE Score of 4 | eSAGE Score of 5 | eSAGE Score of 6 | eSAGE Score of 7 | eSAGE Score of 8 | eSAGE Score of 9 | eSAGE Score of 10 | eSAGE Score of 11 | eSAGE Score of 12 | eSAGE Score of 13 | eSAGE Score of 14 | eSAGE Score of 15 | eSAGE Score of 16 | eSAGE Score of 17 | eSAGE Score of 18 | eSAGE Score of 19 | eSAGE Score of 20 | eSAGE Score of 21 | eSAGE Score of 22
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/4 | 0/1 | 0/2 | 0/4 | 0/6 | 0/2 | 0/2 | 0/3 | 0/4 | 0/5 | 0/5 | 0/8 | 0/6 | 0/3 | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/4 | 0/1 | 0/2 | 0/4 | 0/6 | 0/2 | 0/2 | 0/3 | 0/4 | 0/5 | 0/5 | 0/8 | 0/6 | 0/3 | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/4 | 0/1 | 0/2 | 0/4 | 0/6 | 0/2 | 0/2 | 0/3 | 0/4 | 0/5 | 0/5 | 0/8 | 0/6 | 0/3 | 0/4 | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
The majority of the subjects were Caucasian and highly educated. Results may be limited based on where the patients were recruited and their range of cognitive abilities. The ADCS-ADL scale was used as self-report in subjects without a study partner.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT02544074/Prot_SAP_000.pdf